CLINICAL TRIAL: NCT05389553
Title: The Association Between Fetal Doppler and Uterine Artery Blood Volume at Term of Pregnancy: A Prospective Observational Study.
Brief Title: Fetal Doppler and Uterine Artery Blood Volume Correlation.
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 0010010/i
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Fetal Doppler; Uterine Blood Flow
Keywords: Doppler; Pregnancy; ultrasound; uterine blood flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at term of pregnancy: We included all full-term pregnancies accepted for delivery that received an accurate ultrasound scan before the birth.
  Pregnant women with antepartum hemorrhage, fetal growth restriction, stillbirths, multiple gestations, or congenital abnormalities were excluded.
  Interventions: Other: Ultrasound exam

INTERVENTIONS:
Other: Ultrasound exam — We included all full-term pregnancies accepted for delivery that received an accurate ultrasound scan before the birth

SUMMARY:
To investigate the relationship between uterine artery blood volume and fetal doppler indices at the delivery.

DETAILED DESCRIPTION:
Introduction: To investigate the relationship between uterine artery blood volume and fetal doppler indices at the delivery.

Materials and Methods: This was a prospective cohort study of 50 nulliparous women booking antenatal care at the University of Campania "Luigi Vanvitelli" between May 2022 and September 2022. All full-term pregnancies accepted for delivery will include. Pregnant women with antepartum haemorrhage, stillbirths, multiple gestations, or congenital abnormalities were excluded. Women underwent a transabdominal ultrasound examination of uterine arteries for measurement of Uterine artery blood volume. Pregnancy outcomes were recorded, and linear regression was used to study the relationship between uterine artery blood volume and fetal Doppler indices. SPSS version 25 (Chicago, IL, USA) was used to code, tabulate, and analyze the data. Quantitative data were analyzed using the student's t-test. Qualitative data were analyzed using the Mann-Whitney test. A statistically significant difference was defined as a p-value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* full-term pregnancies (37-42 weeks)

Exclusion Criteria:

* antepartum hemorrhage, fetal growth restriction, stillbirths, multiple gestations, or congenital abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Full-term pregnancies (37-42 weeks) comprised all pregnant women who would give birth at our hospital.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
We estimate the uterine volume and its correlation with the fetal doppler indices | 1 day
  The volume of the uterine arteries will be measured using a doppler ultrasound. We shall also estimate the fetal doppler indices.
  Linear regression will be used to test for a possible relationship between uterus volume blood flow and fetal doppler parameters. Before the delivery, all of these variables will be estimated using an ultrasound exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: No